CLINICAL TRIAL: NCT04557540
Title: Comparison of Intermittent Fasting With Continuous Caloric Reduction in Black Adults of Faith
Brief Title: Weight Loss Interventions for Black Adults of Faith
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 684220; NCI-2020-06640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 684220 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-09-09; First posted 2020-09-21 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Obesity-Related Malignant Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Fasting WORD) (Experimental): Participants receive the Fasting WORD intermittent fasting weight loss intervention consisting of 16 small-group lessons over 1.5 hours each QW for 2 months and then Q2W for 4 months.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Short-Term Fasting
- Arm II (The WORD) (Experimental): Participants receive The WORD CER weight loss intervention consisting of 16 small-group lessons over 1.5 hours each QW for 2 months and then Q2W for 4 months.
  Interventions: Behavioral: Lifestyle Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Lifestyle Therapy — Receive The WORD lifestyle CER weight loss intervention
  Arms: Arm II (The WORD)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Short-Term Fasting — Receive Fasting WORD intermittent fasting weight loss intervention
  Other Names: Intermittent Fasting; Short-term Intermittent Fasting
  Arms: Arm I (Fasting WORD)

SUMMARY:
This trial compares the effect of intermittent fasting versus continuous caloric reduction for the reduction of body weight in Black adults of faith. Intermittent fasting and continuous caloric reduction interventions may help Black adults of faith lose weight, improve their health, and help reduce cancer risk.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Partner with the First Ladies of Western New York (FLOW) to engage 10 community stakeholders from Black churches in the Roswell Park Catchment area in a four-stage process involving information gathering, discussion groups, and mock intervention delivery to create Fasting WORD for Black adults of faith.

II. Implement and determine the initial comparative effectiveness of Fasting WORD with The WORD to reduce body weight, and biomarkers of obesity, inflammation, insulin, and insulin resistance.

SECONDARY OBJECTIVES:

I. Examine the interventions' effects on diet and physical activity. II. Examine participants' adherence and satisfaction with both interventions.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive the Fasting WORD intermittent fasting weight loss intervention consisting of 16 small-group lessons over 1.5 hours each once a week (QW) for 2 months and then once every 2 weeks (Q2W) for 4 months.

ARM II: Participants receive The WORD continuous energy restriction (CER) weight loss intervention consisting of 16 small-group lessons over 1.5 hours each QW for 2 months and then Q2W for 4 months.

After completion of study, participants are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black
* Body mass index (BMI) > 25 kg/m^2
* Associated with a participating church through membership or participation in a church activity
* Cleared by a Primary Care Provider (PCP-Doctor) to be a part of the study
* Not currently on weight loss medications
* Not pregnant or lactating
* Has not lost at least 10% of their body weight in the last 6 months
* Has not had bariatric surgery in the last 10 years
* Able to walk unassisted and continuously for 10 minutes

Exclusion Criteria:

* Adults unable to consent
* Adults unable to complete study measures in English
* Individuals who are not yet adults (infants, children, teenagers)
* Individuals who are pregnant or lactating
* Adults who have had a myocardial infarction (heart attack) or stroke without medical clearance from their primary care physician to participate in the study
* Adults who currently have type 1 or type 2 diabetes without medical clearance from their primary care physician to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Up to 6 months
Changes in body composition | up to 6 months
Change in height | up to 6 months
Change in heart rate | Up to 6 months
Change in blood pressure | AT 6 months
Change in waist circumference | Up to t 6 months
Change in hip circumference | Up to 6 months

SECONDARY OUTCOMES:
Dietary intake | Up to 6 months
  Dietary intake will be assessed by the interview-administered Nutrition Data System for Research (NDSR).
Obesity-related biomarker analysis | Up to 6 months
  Will measure biomarkers related to , including C-peptide, as a marker of insulin secretion Will assay for 6 adipokines including leptin, adiponectin, adipsin, lipocalin-2/NGAL, resistin, and PAI-1 (total) as markers of adiposity and adiposity-related metabolic dysfunction, including insulin resistance, and CRP as a well-characterized and validated marker for systemic inflammation.
glucose metabolism | UP to 6 months
  Change from baseline
changes in Adipokine levels | Up to 6 months
  blood concentration measure
C-Peptide level | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeary, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States